CLINICAL TRIAL: NCT05520359
Title: Transcutaneous Stimulation and Mobility Device Use for Individuals With Neurologic Conditions
Brief Title: Spinal Stimulation and Mobility Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Katherine Steele, Professor, Mechanical Engineering, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00014877
Record Dates: First submitted 2022-08-22; First posted 2022-08-29 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cerebral Palsy; Stroke; Premature Birth; Hypoxic-Ischemic Encephalopathy; Periventricular Leukomalacia
Keywords: Pediatric; Mobility Aids; Assistive Technology; Spinal Stimulation
MeSH Terms: conditions — Cerebral Palsy; Stroke; Premature Birth; Hypoxia-Ischemia, Brain; Leukomalacia, Periventricular | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized order of visits with individual and combined effects of mobility devices and spinal stimulation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Neurologic Disorders (Experimental): Evaluation of individual and combined effects of mobility devices and spinal stimulation for individuals with neurologic disorders.
  Interventions: Device: Mobility Device; Device: Spinal Stimulation

INTERVENTIONS:
Device: Mobility Device — Use of mobility device during session.
  Other Names: Biomotum SPARK; Trexo; Portable Mobility Aid for Children (PUMA, ENLITEN)
Device: Spinal Stimulation — A stimulator will be used non-invasively stimulate the spine at the neck and/or lower back (cervical and/or lum
  Other Names: SpineX

SUMMARY:
This research study will combine non-invasive spinal stimulation with mobility devices to examine the acute impact of the individual and combined effects of these innovative techniques on mobility in children with cerebral palsy.

DETAILED DESCRIPTION:
For people with neurological conditions, excessive and inappropriate muscle activity resulting from injured sensory pathways (e.g., spasticity or hypertonicity) contributes to inefficient movement, bone deformities, pain, and other comorbidities. Research with humans and animals have highlighted the critical importance of both motor and sensory pathways for motor learning after neurologic injury. However, the best techniques for engaging motor and sensory pathways in a way that brings high quality mobility are not well understood. With this study we will examinee how increased sensory feedback, through mobility device use and electrical spinal stimulation, impact movement mechanics in people with neurological conditions to inform long-term studies and eventual implementation into clinical practice.

Mobility devices offer a promising approach to improve mobility rehabilitation through engagement of sensory and motor pathways. These devices can either assist in movement by providing support to perform an activity or they can be used to provide resistance to build strength. Mechanistically how these devices impact movement mechanics is still not well understood.

Electrical spinal stimulation with intensive, repetitive training has demonstrated exciting potential to improve limb function after neurologic injury. Spinal stimulation has shown to improve motor function with long-term training. Stimulation is hypothesized to improve motor pathways through boosting sensory input. However, the neuromechanical effects of stimulation as a result of increased sensory feedback over an acute time frame has not been explored in efforts to test this hypothesis.

This study aims to evaluate the acute effects of increased afferent feedback in individuals with neurological conditions via mobility devices and spinal stimulation. Understanding how these approaches affect the quantity and quality of movement in the short term is a first step before determining potential treatment outcomes. In this research, we will quantify the neuromechanics of movement with and without these approaches for individuals with neurologic disorders.

ELIGIBILITY:
Inclusion Criteria:

* have a neurologic condition
* are 4-70 years of age
* have stable medical condition
* can perform simple cued motor tasks and who can follow 2-3 step commands
* who are volunteering to be involved in this study
* can provide feedback on comfort and experience during lab visits

Exclusion Criteria:

* have significant medical disease; including uncontrolled systemic hypertension with values above 170/100 mmHg; cardiac or pulmonary disease; uncorrected coagulation abnormalities or need for therapeutic anticoagulation.
* have cardiovascular or musculoskeletal disease or injury that would prevent full participation in physical therapy intervention
* have a history of uncontrolled seizures
* have unhealed fracture or other musculoskeletal impairment that might interfere with lower extremity rehabilitation or testing activities
* are dependent on ventilation support
* have implanted stimulator (e.g. epidural stimulator, vagus nerve stimulator, pacemaker, cochlear implant, etc) or drug delivery device (e.g. baclofen pump)
* have history of orthopedic surgery in lower extremities or neurosurgery that may be a confounding factor for interpretation of the results (such as tendon transfer, tendon or muscle lengthening for spasticity management, injection therapies to lower extremity muscles, etc.) in last 12 months
* have established osteoporosis and taking medication for osteoporosis treatment.
* have rheumatic diseases (rheumatoid arthritis, systemic lupus erythematosus, etc.)
* have active cancer

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08-04 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Coordination | Comparing first and last minute of walking on treadmill at each experimental session.
  Change in level of co-contraction between the plantarflexor and tibialis anterior muscles during the gait cycle monitored from electromyography recordings.

SECONDARY OUTCOMES:
Modified Ashworth Scale | Physical exam conducted at the beginning and end of each experimental session.
  Change in summed score of spasticity from lower-extremity muscles. Lower values indicate less spasticity.
Plantarflexor Muscle Strength | Physical exam conducted at the beginning and end of experimental session.
  Change in maximum voluntary contraction level of the plantarflexor muscles taken as the average of three trials where the participant exerts the maximum amount of force measured from a handheld dynamometer with verbal encouragement.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Steele, PHD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No